CLINICAL TRIAL: NCT05993598
Title: The Effect of Hippotherapy Applied on Different Sitting Surfaces on Sitting Balance and Walking Speed in Children With Special Needs
Brief Title: The Effect of Hippotherapy Applied on Different Seating Surfaces in Children With Special Needs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medipol University Hospital (Other)
Responsible Party: Principal Investigator, Ebru Sever, PhD, PT, Istanbul Medipol University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BURAKEMİRHAN
Record Dates: First submitted 2023-07-31; First posted 2023-08-15 (Actual); Last update posted 2023-08-15 (Actual); Status verified 2023-08

CONDITIONS: Special Needs Children
Keywords: hippotherapy; sitting balance; child with special needs; walking speed
MeSH Terms: interventions — Equine-Assisted Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1 (Saddled) (Experimental): Each group did a 30-minute hippotherapy session in the manege area. Before the application, the sitting balance of the children was evaluated by playing the Nintendo Wii Balance Platform and the Basic Balance Game. In addition, 10 m walking test was applied for walking speed. These assessments were repeated after the 30-minute session.
  Interventions: Other: hippotherapy
- Group 2 (Saddleless, direct contact with horse) (Experimental): Each group did a 30-minute hippotherapy session in the manege area. Before the application, the sitting balance of the children was evaluated by playing the Nintendo Wii Balance Platform and the Basic Balance Game. In addition, 10 m walking test was applied for walking speed. These assessments were repeated after the 30-minute session.
  Interventions: Other: hippotherapy
- Group 3 (Different tissue to be put on the saddle) (Experimental): Bubbled nylon (pat-to-pat) was used as a different texture. Each group did a 30-minute hippotherapy session in the manege area. Before the application, the sitting balance of the children was evaluated by playing the Nintendo Wii Balance Platform and the Basic Balance Game. In addition, 10 m walking test was applied for walking speed. These assessments were repeated after the 30-minute session.
  Interventions: Other: hippotherapy

INTERVENTIONS:
Other: hippotherapy — Evaluation parameters were applied to 30 children with special needs at the beginning of the session. After the evaluation, each group was given a 30-minute hippotherapy session in the manege area. During the practice, the child simply sat on the horse. The horse was asked to maintain its balance by adapting to the oscillations it creates while walking on the sand. Immediately after the 30-minute application, the initial evaluations were made again. As a result, it was investigated whether hippotherapy applied on different sitting surfaces in children with special needs had an effect on sitting balance and walking speed.

SUMMARY:
The effect of hippotherapy, which will be applied to children with special needs in a single session, on sitting balance and walking speed under the supervision of a physiotherapist was investigated. 30 randomly selected children with special needs between the ages of 3-18 who were referred to the Gebze Equestrian Training Center were included in the study. The children were randomly divided into 3 groups: 10 in the saddle, 10 naked (direct contact with the horse), and 10 in the hippotherapy group, in which a cloth of different texture was placed on the horse. Each group did a 30-minute hippotherapy session in the manege area. Before the application, the sitting balance of the children was evaluated by playing the Nintendo Wii Balance Platform and the Basic Balance Game. In addition, 10 m walking test was applied for walking speed. These assessments were repeated after the 30-minute session. It was checked whether the application had an effect on balance and walking speed. Comparisons between the groups were made and it was examined which application was more effective on balance and walking speed.

ELIGIBILITY:
Inclusion Criteria:

* Having a child with special needs between the ages of 3-18,
* Children with a diagnosis of Cerebral Palsy (CP) have a level of 1 and 2 according to the Gross Motor Function Classification System,
* Ability to understand simple commands,
* Ability to sit unaided for at least 10 seconds,

Exclusion Criteria:

* Presence of clinical conditions that may pose an obstacle
* Lack of cooperation
* Presence in another study performed at the same time as the study
* Lack of family approval.

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Actual)
Dates: Start 2023-01-17 (Actual); Primary Completion 2023-02-17 (Actual); Study Completion 2023-05-10 (Actual)

PRIMARY OUTCOMES:
BeCure Balance Evaluation System | 11 weeks
  BeCure Balance Assessment System protocol; It was planned to determine the amount of change in the center of gravity in the x and y axes and the position of the body center of gravity during balancing by sitting on the board for 30 seconds with eyes open, with images.

SECONDARY OUTCOMES:
Ten(10) Meter Walking Test(sec) | 11 weeks
  In this test, the person is asked to walk at their own normal pace in a pre-measured 10 meter area (if using walking aid, it will be done with it). The time starts when the person's foot is on the starting line and ends when they cross the finish line. Two measurements are made and the best value is recorded in meters per second (m/s).
Gross Motor Function Classification System (GMFCS) | 11 weeks
  It was used to evaluate the motor functions of participants with a diagnosis of cerebral palsy. It is a standardized method that classifies motor function differences in sitting and walking at 5 levels. If we examine the 5 levels; Level I walks without restrictions; Level II walks with restrictions; Level III walks using hand-held mobility devices; Level IV, independent self-mobility is limited and may use a motorized mobility vehicle; Level V is transported in a manual wheelchair.

CONTACTS AND LOCATIONS:
Overall Officials: Ebru SEVER, Lecturer, Study Director — Department of Physiotherapy & Rehabilitation
Locations (1):
- Gebze Municipality Equestrian Training Center, Kocaeli, Gebze, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No